CLINICAL TRIAL: NCT04439981
Title: Beneficial Effect of Curcuma Extract In Muscle Damage (Study in Soccer Athlete): Randomized Clinical Trial
Brief Title: Curcuma Extract Beneficial for Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Semarang (Other)
Responsible Party: Principal Investigator, Ali Rosidi, Dr, Dean of Faculty of Nursing and Health, Universitas Muhammadiyah Semarang, Universitas Muhammadiyah Semarang
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Curcuma
Record Dates: First submitted 2020-06-11; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Athletes Foot
Keywords: Curcuma extract; ice cream; inflammation; muscle damage
MeSH Terms: conditions — Tinea Pedis; Inflammation | interventions — Ice Cream

STUDY DESIGN:
Intervention Model Description: Subjects were divided by 2 groups: control group (n=10), treated by ice cream without any Curcuma extract supplementation; and treatment group (n=10), treated by ice cream supplemented by Curcuma extract.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): treated by ice cream without any Curcuma extract supplementation
  Interventions: Dietary Supplement: Ice cream
- Treatment Group (Experimental): treated by ice cream supplemented by Curcuma extract
  Interventions: Dietary Supplement: Ice cream

INTERVENTIONS:
Dietary Supplement: Ice cream — Curcumin extract was added into ice cream

SUMMARY:
Muscle damage and inflammation is a clinical problem caused by the unimpeachable body adaptation of strenuous exercise through increasing free radicals. Antioxidants content in Curcuma is hypothesized to alleviate the free radicals. This study aimed to examine the effect of Curcuma extract in the form of ice cream to improve muscle damage and inflammation of soccer athletes caused by strenuous exercise. This study was experimental study with pre-post control group design. Male soccer athlete (n=20) were divided into treatment group (n=10) and control group (n=10). The treatment group was treated by Curcuma extract ice cream for 21 days. Blood samples of creatine kinase (as muscle damage marker) and IL-6 (as inflammation marker) were quantified.

DETAILED DESCRIPTION:
Muscle damage is a clinical problem caused by the adaptation process in strenuous exercise of soccer athletes which free radical is the main culprit of the damage. There is a significant increment of muscle damage after strength exercise using leg press. Physical exercise leads to inflammation process in endothelial cells of blood vessel which can be marked by releasing cytokine. Interleukin-6 (IL-6) is one of cytokine pro-inflammation and this marker is used as an indicator for inflammation of micro-trauma in muscle during strenuous exercise.

Normally, free radical generation will be stabilized by endogenous antioxidant secretion such as superoxide dismutase (SOD), glutathione peroxidase (GPx), and catalase; nevertheless, body needs exogenous antioxidant to support endogenous antioxidant as a scavenger of free radical in such condition.

Muscle damage due to the strenuous exercise should be managed to avoid the pain feeling and subsequently decrease athlete performances. Some previous studies used herbs such as ginger (Zingiber officinale), ginseng (Panax quinquefolium), and Curcuma to relieve the muscle damage and inflammation resulting from high-intensity exercise.The Curcuma extract treatment to the athlete gained lack of success; therefore, supplementation to food products might use to increase acceptability. Ice cream is one of the products, which has a broad segment market and every single person regardless of age is fond of it.

Curcumin is an antioxidant substance contained in Curcuma and it has better antioxidant capacity compared to the other component in Curcuma such as demetoksicurcumin and bisdemetoksicurcumin.Besides, curcumin has an efficient reaction with superoxide radicals as well as lipid antioxidants has, and the reaction leads to superoxide catalytic degradation in which curcumin represents as a superoxide dismutase. This study aimed to examine the Curcuma extract effect which has been supplemented to own-made ice cream in muscle damage and inflammation of soccer athletes after having strenuous exercise.

ELIGIBILITY:
Inclusion Criteria:

* male
* 14-18 year-old
* does not have an acute and chronic
* hemoglobin level ≥13 g/L
* nutrition status normal (BMI >18.5-25.0)
* no coffee consumption
* no alcohol consumption
* no drugs consumption
* no smoking
* no vitamin and other supplements consumption at least two weeks before this study was conducted
* no additional exercise except the programmed exercise

Exclusion Criteria:

* Subject did not comply the procedure of the study

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Lactic acid change | 21 days
  Change from baseline lactic acid at 21 days taken in the lab from venous blood specimen using spectrophotometric method
Hemoglobin change | 21 days
  Change from baseline hemoglobin at 21 days taken in the lab from venous blood specimen using cyanmethemoglobin method
IL-6 change | 21 days
  Change from baseline IL-6 at 21 days taken in the lab from venous blood specimen using ELISA method
Creatinine kinase change | 21 days
  Change from baseline creatinine kinase at 21 days taken in the lab from venous blood specimen using ELISA method

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rosidi, Doctor, Principal Investigator — Universitas Muhammadiyah Semarang
Locations (1):
- Badan Pusat Pendidikan dan Pelatihan Olahraga Pelajar (BPPLOP) Semarang, Indonesia, Semarang, Provinsi, Indonesia

IPD SHARING:
Plan to Share IPD: No